CLINICAL TRIAL: NCT00848172
Title: Double-Blind, Placebo Controlled Pilot-Study of Octanoic Acid in Essential Tremor
Brief Title: Double-Blind, Placebo Controlled Pilot Study of Octanoic Acid in Essential Tremor
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Mark Hallett, Chief, Human Motor Control Section, National Institute of Neurological Disorders and Stroke (NINDS)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 090084; 09-N-0084
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Results first posted 2012-12-27 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-11

CONDITIONS: Essential Tremor
Keywords: Essential Tremor; Octanol; Octanoic Acid; Ethanol; Accelerometry
MeSH Terms: conditions — Essential Tremor | interventions — octanoic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Octanoic Acid (Active Comparator)
  Interventions: Drug: Octanoic Acid
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Octanoic Acid — 4mg/kg
  Arms: Octanoic Acid
Drug: Placebo — identical capsules
  Arms: Placebo

SUMMARY:
Background:

* Essential tremor (ET) is a neurological disorder characterized by uncontrollable shaking. Several medications are used to treat ET; however, they are often only partly effective and can have side effects.
* Research studies have shown that octanol, a food additive similar to alcohol, can improve tremor in animals. Octanol is less likely to make people drunk than alcohol. Two earlier NIH studies found that one form of octanol, called 1-octanol, did improve tremor in some people and had few side effects.
* In the body, 1-octanol is converted to octanoic acid. Researchers are interested in finding out whether octanoic acid can help people with ET.

Objectives:

* To find out if octanoic acid can improve hand tremor in people with essential tremor.
* To measure levels of octanoic acid in the blood after it is taken.

Eligibility:

* Patients 21 years of age and older with ET, who are willing to abstain from alcohol, caffeine, and all medications as required by the study and who are willing and able to fast for up to 12 hours at a time.
* Participants may not be of Asian or Native American ancestry because of genetic susceptibilities to the intoxicating effects of the study drug.

Design:

* This study requires a 3-day hospital admission as well as two outpatient visits.
* Visit 1 (outpatient): Screening visit and blood alcohol level test
* Medical history, physical and neurological examination, a blood test, and an electrocardiogram to measure heart function. Women who are able to get pregnant will have a urine pregnancy test.
* Patients will consume 1.5 ounces of alcohol per drink (up to three drinks at least 30 minutes apart), and be tested to evaluate how the tremor responds. Researchers will draw blood to measure blood alcohol level about 1 hour after the first drink and closely monitor patients for signs of intoxication.
* Inpatient examination
* Preparation: Researchers will prepare a schedule to stop any tremor medications that patients might be on. Patients may not drink alcohol or eat or drink anything with caffeine, including chocolate, for at least 2 days before admission.
* Day 1: Vital signs, blood (and urine pregnancy) tests, and electrocardiogram. Patients will be asked to wear a tremor monitor, similar to a wristwatch. Patients will also have IV lines inserted for blood draws.
* Days 2 and 3: Randomized study medication (octanoic acid on one day, placebo on the other day). Patients will fast before taking the drug, but will be allowed to eat and drink after the tests are completed (around noon).
* Blood will be drawn before taking the study drug and again (a total of nine times) after taking the drug.
* Tremor will be measured during the study, before and after taking the drug.
* Visit 2 (outpatient): 4 to 7 days after discharge
* Blood test and an electrocardiogram, and a series of questionnaires regarding the study.

DETAILED DESCRIPTION:
OBJECTIVE:

We propose a study to examine the safety and efficacy of octanoic acid in essential tremor (ET).

STUDY POPULATION:

We will study 19 adult subjects with ethanol-responsive ET.

DESIGN:

Octanoic acid will be tested in a double-blind, randomized, placebo-controlled, cross-over design in 19 patients with essential tremor. The active study medication and placebo will be administered as oral single morning doses on consecutive days in a randomized sequence. All subjects will receive a dose that was defined as being safe according to available toxicity data (4mg/kg) and will be monitored closely during the total inpatient study phase of three days (day 0: baseline; days 1-2: active study days).

OUTCOME MEASURES:

The primary outcome measure for this study will be the effect on tremor power of the dominant hand, 80 minutes after administration of the study substance, compared to placebo. Tremor power will be measured using accelerometry with loading to test central tremor component. Secondary outcome measures include recordings of tremor power as measured by accelerometry at multiple other time points up to 300 min after administration, also recorded from the non-dominant hand and without loading. The change in tremor severity documented by spirography and actigraphy as well as data collected regarding drug safety (laboratory testing, documentation of vital signs, adverse events questionnaire and intoxication scale) as well as the pharmacokinetic and pharmacodynamic properties will act as further secondary outcome parameters.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Male or female patients with alcohol-responsive ET according to published clinical criteria
* Tremor in both upper limbs should be predominant feature of ET
* Subjects must be willing and safely able to comply with the study protocol and therefore abstain from any medication for the treatment of tremor for a period of at least 5 plasma half-lives of the individual drug prior to study participation. (For Propranolol/Inderal(Registered Trademark), Gabapentin/Neurontin(Registered Trademark), Topiramate/Topamax(Registered Trademark) this will be 4 days; for Primidone/Mysoline(Registered Trademark): 28 days).
* Subjects must be willing to refrain from alcohol and caffeine intake starting 48 hr prior to hospitalization until study termination
* Subject must be willing and able to fast for periods of up to 12 hours during the study

EXCLUSION CRITERIA:

* Patients with any other significant pathological finding in the neurological examination other than typical symptoms of ET
* Acute or chronic severe medical conditions which would preclude the subject from participating (e.g., severe heart disease NYHA grade 3 or 4, renal failure, hepatic failure, lung disease, uncontrolled hyperthyroidism)
* Subjects with diabetes mellitus, hypoglycemia or severe hyperlipidemia (must be documented by referring physician with copy of last fasting routine blood test within one year before the screening visit including glucose and lipid levels; according to NIH guidelines, fasting LDL levels of greater than or equal to 160 mg/dl are considered severe hyperlipidemia; if under treatment, LDL-levels less than 160 have to be documented to be eligible for the study)
* Subjects with active or past alcohol abuse or dependence
* Subjects with concomitant therapy with warfarin or NSAIDs, when taken on a regular basis and cannot be discontinued at least 14 days prior to study participation, because of potential interactions with octanoic acid (displacement of albumin binding in human serum)
* Subjects with clinically significant abnormalities on their baseline laboratory tests
* Subjects aged less than 21 years
* Female subjects who are pregnant or lactating
* Subjects with cognitive impairment interfering with the ability to give informed consent or to cooperate during the study
* Subjects of Far East Asian or Native American descent, who may possess variant alleles of the genes for alcohol metabolism, i.e., alcohol dehydrogenase and aldehyde dehydrogenase, resulting in altered (slower) metabolism and potentially increased sensitivity to alcohols and their metabolites
* Subjects where no written informed consent is received or subjects who are unwilling to cooperate during the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Zesiewicz TA, Elble R, Louis ED, Hauser RA, Sullivan KL, Dewey RB Jr, Ondo WG, Gronseth GS, Weiner WJ; Quality Standards Subcommittee of the American Academy of Neurology. Practice parameter: therapies for essential tremor [RETIRED]: report of the Quality Standards Subcommittee of the American Academy of Neurology. Neurology. 2005 Jun 28;64(12):2008-20. doi: 10.1212/01.WNL.0000163769.28552.CD. Epub 2005 Jun 22. PMID 15972843
- [Background] Louis ED, Barnes L, Albert SM, Cote L, Schneier FR, Pullman SL, Yu Q. Correlates of functional disability in essential tremor. Mov Disord. 2001 Sep;16(5):914-20. doi: 10.1002/mds.1184. PMID 11746622
- [Background] Stolze H, Petersen G, Raethjen J, Wenzelburger R, Deuschl G. The gait disorder of advanced essential tremor. Brain. 2001 Nov;124(Pt 11):2278-86. doi: 10.1093/brain/124.11.2278. PMID 11673328

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with a diagnosis of ET were recruited by referral from the Motor Control outpatient clinic, a listing on the NINDS web page, and from the general community.
Pre-assignment Details: 29 subjects (12f, 17m) were screened for eligibility. 10 subjects were considered screening failures due to the following reasons: failure to confirm ET according to diagnostic consensus criteria (n=7), other medical conditions precluding a safe participation (n=2), or the lack of objective alcohol-response (n=1). Nineteen subjects were randomized.
Groups:
- Sequence OA / Placebo: During the 3-day inpatient Visit 2 (Drug Administration), after the admissions day (day 1 of Visit 2) patients randomized to Sequence OA / Placebo received a single oral dose of 4 mg/kg OA on the second day of Visit 2, and matching Placebo on the third day of Visit 2. Patients were discharged at the end of the third day of Visit 2, which ended this study visit.
- Sequence Placebo / OA: During the 3-day inpatient Visit 2 (Drug Administration), after the admissions day (day 1 of Visit 2) patients randomized to Sequence OA / Placebo received Placebo on the second day of Visit 2, and a single oral dose of 4 mg/kg OA on the third day of Visit 2. Patients were discharged at the end of the third day of Visit 2, which ended this study visit.
Period: Visit 2 - Drug Administration
Arm/Group | Sequence OA / Placebo | Sequence Placebo / OA
Started | 10 | 9
Completed | 10 | 8
Not Completed | 0 | 1
Period: Visit 3 - Follow Up
Arm/Group | Sequence OA / Placebo | Sequence Placebo / OA
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sequence OA / Placebo: First day: octanoic acid Second day: placebo
- Sequence Placebo / OA: First day: placebo Second day: octanoic acid
- Total: Total of all reporting groups
Arm/Group | Sequence OA / Placebo | Sequence Placebo / OA | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 4 | 10
  >=65 years | 4 | 5 | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 59.90 (10.97) | 64.22 (8.60) | 61.95 (9.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 6 | 8 | 14
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Normalized Accelerometric Tremor Power, Dominant Hand, 80min After Administration, Weighted Condition
Description: Postural tremor was measured using accelerometry with a motion sensor (accelerometer) placed at the dorsum of each hand, and tremor recorded simultaneously with surface-electromyography of wrist flexors and extensors for 2 minutes at each time-point. The recording was repeated with 1 lbs weight added to each wrist, which was described to record the central tremor component. The primary outcome measure was defined as tremor power of the central tremor component (after the addition of weight) 80 minutes after administration, measured at the dominant hand, normalized to baseline (baseline = 1), and comparing octanoic acid vs. placebo. Ratio of tremor power at 80 min divided by tremor power at baseline used for outcome measure calculation.
Time Frame: 80 min after administration of the study drug on day 1 and 2 of Visit 2
Population: 2 patients were excluded from primary outcome measure analysis because of one subject was withdrawn prior to drug administration due to an SAE, and one subject did not exhibit a central tremor component (primary measure), on the day of administration.
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Octanoic Acid | Placebo
Number analyzed (Participants) | 17 | 17
ratio | 0.669 [0.489 to 1.548] | 0.798 [0.540 to 1.342]
Statistical Analysis 1: Comparison: Octanoic Acid vs Placebo; Test type: Superiority or Other; p = 0.345, Mixed Models Analysis

2. Secondary Outcome: Normalized Tremor Power, 300 Min After Administration, Weighted Condition, Dominant Hand, OA vs Placebo
Description: As described at the section for the primary outcome, normalized accelerometric tremor accelerometry was measured at other time-points to describe a time-course of effect. This stated secondary outcome compared normalized (baseline = 1) accelerometric at the last time-point 300 min post dose after OA vs Placebo. Ratios of tremor power at 300 min divided by tremor power at baseline used for outcome measure calculation.
Time Frame: 300 min post dose
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Octanoic Acid | Placebo
Number analyzed (Participants) | 17 | 17
ratio | 0.689 [0.506 to 1.111] | 1.071 [0.542 to 1.995]
Statistical Analysis 1: Comparison: Octanoic Acid vs Placebo; Test type: Superiority or Other; p = 0.031, Mixed Models Analysis

3. Secondary Outcome: TMax Octanoic Acid
Description: Time to plasma peak OA
Time Frame: between 5 and 300 min post dose
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Octanoic Acid Tmax
Number analyzed (Participants) | 18
min | 72.8 (34.3)

4. Secondary Outcome: PK: AUC After OA
Description: Area under the curve of PA plasma levels after administration
Time Frame: 5 to 300 min post dose
Measure: Mean (Standard Deviation); unit: hr*ng/ml
Arm/Group | Octanoic Acid AUC
Number analyzed (Participants) | 18
hr*ng/ml | 1860.9 (474.7)

ADVERSE EVENTS:
Groups:
- Non-drug Related: AE was considered to be non-drug related, if no temporal connection was present between AE occurrence and drug administration (e.g. if AE occurred during the study, but prior to drug-administration), or an AE was clearly related to a study procedure (e.g. PICC line) rather than the study drug.
Arm/Group | Octanoic Acid | Placebo | Non-drug Related
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19 | 2/19
Other Adverse Events (participants affected / at risk) | 7/18 | 7/19 | 4/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Octanoic Acid (N=18) | Placebo (N=19) | Non-drug Related (N=19)
Troponin I elevation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Patient with food-borne illness with consecutive Troponin I elevation before OA administration
bleeding from PICC insertion site (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) — Patient who (contrary to instructions given) removed pressure dressing on PICC insertion site after line-removal at the end of visit 2, who consecutively experienced mild bleeding. After re-application of pressure dressing, bleeding stopped.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Octanoic Acid (N=18) | Placebo (N=19) | Non-drug Related (N=19)
Fatigue (General disorders) | 3 (3) | 2 (2) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Pain at PICC insertion site (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Dry Mouth (General disorders) | 0 (0) | 1 (1) | 1 (1)
Taste Change (General disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No